CLINICAL TRIAL: NCT02935894
Title: Investigating the Stability, Variability and Mechanism of Incorporation of Lipid Mediators Into Eccrine Sweat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 929370
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-04

CONDITIONS: Stability & Variability of Lipid-derived Molecules in Sweat
Keywords: oxygenated lipids; metabolic profiling; sphingoid bases; ceramides; endocannabinoids; non-invasive sampling
MeSH Terms: interventions — Ibuprofen; Exercise; Pilocarpine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group (Experimental): All subjects will participate in 4 study day visits in the same order.
  1. compare sweat collected following pharmacological stimulation of sweating (using the drug pilocarpine) to sweat collected following physiological induction of sweating (exercise using a stationary bicycle).
  2. compare sweat collected following stimulation of sweating by the drug pilocarpine from the inner part of the forearm (near the wrist) to upper surface of thigh (near the knee).
  3. collect sweat following stimulation of sweating by the drug pilocarpine from the inner part of both forearms (near the wrist).
  4. collect blood and sweat samples before and 30 minutes, 2 hours and 4 hours after consumption of 400 mg of ibuprofen.
  Interventions: Drug: Ibuprofen; Other: Physiological induction of sweating; Drug: Pilocarpine

INTERVENTIONS:
Drug: Ibuprofen — 400 mg ibuprofen given to inhibit cyclooxygenase metabolism
Other: Physiological induction of sweating — 15 minutes exercise at 60-80% oxygen consumption to induce sweating
  Other Names: Exercise
Drug: Pilocarpine — Iontophoresis with a 1.5 milliampere (mA) current using a gel disc containing a 5% pilocarpine nitrate solution to induce sweating
  Other Names: Pilogel

SUMMARY:
The purpose of this study is to see what the differences are in sweat (amount and small molecule content) collected from different sites of the body and by different methods of sweat stimulation. Additionally, the investigators want to know whether the amount and small molecule content of the sweat is the same in an individual over time, and the same across individuals at a given time. Finally, the investigators want to know how consumption of over-the-counter anti-inflammatory drugs such as ibuprofen will affect the inflammatory mediator content of sweat and how that compares to blood. This information will help to better understand the composition and behavior of sweat and assess its potential utility as a routine clinical tool in skin research.

DETAILED DESCRIPTION:
Subjects will participate in 4 study day visits that will be scheduled about 1- week apart. During the first study visit, the investigators will compare sweat collected following pharmacological stimulation of sweating (using the drug pilocarpine) to sweat collected following physiological stimulation of sweating (using a stationary bicycle). During the second study visit, the investigators will collect sweat following stimulation of sweating by the drug pilocarpine from the inner part of the forearm (near the wrist) and also the upper surface of the thigh (near the knee). During the third study visit, the investigators will collect sweat following stimulation of sweating by the drug pilocarpine from the inner part of both forearms (near the wrist). During the fourth study visit, the investigators will collect a sweat sample following stimulation of sweating by the drug pilocarpine from the inner part of the forearm (near the wrist) and a blood sample (about one teaspoon) from the other arm. After blood and sweat collection, participants will consume 400 mg (two tablets) of ibuprofen. The investigators will then collect blood and sweat from 30 minutes, 2 hours and 4 hours after participants consume the ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 y
* Male
* Weight > 110 pounds

Exclusion Criteria:

* Diagnosed active chronic diseases for which the individual is currently taking daily medication, including but not limited to:

  * Diabetes mellitus
  * Cardiovascular disease
  * Cancer
  * Gastrointestinal disorders
  * Kidney disease
  * Liver disease
  * Bleeding disorders
  * Asthma
  * Autoimmune disorders
  * Hypertension
  * Osteoporosis
* Recent minor surgery (within 4 wk) or major surgery (within 16 wk)
* Recent antibiotic therapy (within 4 wk)
* Recent hospitalization (within 4 wk)
* Use of over-the-counter or prescription medications at the time of the study that directly affect endpoints of interest (e.g. hyperlipidemia, glycemic control, steroids, statins, anti-inflammatory agents, and weight loss aids)
* Adults who are not able to consent
* Under current medical supervision
* Ibuprofen intolerance or allergy
* Those with a bleeding disorder
* Current enrollee in a clinical research study.
* Individuals with blood clotting or platelet defect disorders
* Individuals with orthopedic limitations or cardiovascular risk that preclude participation in the physiological stimulation of sweat by light exercise portion of the study
* Individuals who are trained athletes or that regularly perform physical activity defined as "vigorous" by the Centers for Disease Control and Prevention

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Newman, Ph.D., Principal Investigator — USDA-ARS-Western Human Nutrition Research Center
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group: Subjects will participate in 4 study visits in the same order.
  1. compare sweat collected following pharmacological stimulation of sweating (using the drug pilocarpine) to sweat collected following physiological induction of sweating (exercise using a stationary bicycle).
  2. compare sweat collected following stimulation of sweating by pilocarpine from the inner part of the forearm (near the wrist) to upper surface of thigh (near the knee).
  3. collect sweat following stimulation of sweating by the drug pilocarpine from the inner part of both forearms (near the wrist).
  4. collect blood and sweat samples before and 30 minutes, 2 hours and 4 hours after consumption of 400 mg of ibuprofen.
  Ibuprofen: 400 mg ibuprofen given to inhibit cyclooxygenase metabolism
  Physiological induction of sweating: 15 minutes exercise at 60-80% oxygen consumption to induce sweating
  Pilocarpine: Iontophoresis with a 1.5 milliampere (mA) current using a gel disc containing a 5% pilocarpine
Period: Overall Study
Arm/Group | Single Group
Started | 14
Completed | 13
Not Completed | 1
Not completed — Subject dismissed | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Group: All subjects will participate in 4 study day visits in the same order.
  1. compare sweat collected following pharmacological stimulation of sweating (using the drug pilocarpine) to sweat collected following physiological induction of sweating (exercise on a stationary bicycle).
  2. compare sweat collected following stimulation of sweating by the drug pilocarpine from the inner part of the forearm (near the wrist) to upper surface of thigh (near the knee).
  3. collect sweat following stimulation of sweating by the drug pilocarpine from the inner part of both forearms (near the wrist).
  4. collect blood and sweat samples before and 30 minutes, 2 hours and 4 hours after consumption of 400 mg of ibuprofen.
  Ibuprofen: 400 mg ibuprofen given to inhibit cyclooxygenase (COX) metabolism
  Physiological induction of sweating: 15 minutes exercise at 60-80% oxygen consumption to induce sweating
  Pilocarpine: Iontophoresis with a 1.5 milliampere (mA) current using a gel disc containing a
Arm/Group | Single Group
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14
Height [Mean (Standard Deviation); unit: centimeters] | 179.2 (6.2)
Weight [Mean (Standard Deviation); unit: kilograms] | 82.6 (15.9)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 25.8 (5.0)
Perceived Exercise Intensity [Mean (Standard Deviation); unit: units on a scale] — Based on Physical Activity Intensity guidelines published by the Centers for Disease Control and Prevention. Intensity is based on an arbitrary scale where 0 = Sedentary, 1 = Light, 2 = Moderate, 3 = Strenuous
  units on a scale | 1.6 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Volar Forearm Sweat Lipid Mediator Concentrations Following Pilocarpine Stimulation
Description: Approximately 150 lipid mediators will be measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Assayed lipid mediators include oxygenated lipids, endocannabinoids and endocannabinoid-like molecules, and sphingolipids.
Time Frame: measured at study visit 1, 2 and 3; detected lipid mediator concentrations for study visit 1 reported
Population: Of the 14 subjects recruited for this study, only 7 provided usable data for this primary outcome.
Measure: Mean (Standard Deviation); unit: picomoles per milliliter
Groups:
- Single Group: All subjects will participate in 4 study day visits in the same order.
  1. compare sweat collected following pharmacological stimulation of sweating (using the drug pilocarpine) to sweat collected following physiological induction of sweating (exercise using a stationary bicycle).
  2. compare sweat collected following stimulation of sweating by the drug pilocarpine from the inner part of the forearm (near the wrist) to upper surface of thigh (near the knee).
  3. collect sweat following stimulation of sweating by the drug pilocarpine from the inner part of both forearms (near the wrist).
  4. collect blood and sweat samples before and 30 minutes, 2 hours and 4 hours after consumption of 400 mg of ibuprofen.
  Ibuprofen: 400 mg ibuprofen given to inhibit COX metabolism
  Physiological induction of sweating: 15 minutes exercise at 60-80% oxygen consumption to induce sweating
  Pilocarpine: Iontophoresis with a 1.5 milliampere (mA) current using a gel disc containing a 5% pilocarpine
Arm/Group | Single Group
Number analyzed (Participants) | 7
picomoles per milliliter
  9-HODE | 20 (9.8)
  13-HODE | 46 (28)
  9-HOTrE | 2.2 (1.2)
  13-HOTrE | 3.5 (1.8)
  5-HETE | 0.1 (0.07)
  8-HETE | 0.23 (0.062)
  9-HETE | 0.12 (0.062)
  11-HETE | 0.15 (0.055)
  12-HETE | 0.85 (0.94)
  15-HETE | 0.43 (0.25)
  12-HEPE | 0.086 (0.044)
  9,10-e-DiHO | 85 (37)
  9,10-DiHOME | 4.4 (3)
  12,13-DiHOME | 3.4 (2.3)
  9,10-DiHODE | 0.85 (1.1)
  12,13-DiHODE | 0.5 (0.31)
  15,16-DiHODE | 2.7 (3.9)
  5,6-DiHETrE | 5.3 (2.5)
  8,9-DiHETrE | 0.73 (0.43)
  11,12-DiHETrE | 0.51 (0.29)
  14,15-DiHETrE | 0.65 (0.4)
  9,10-EpOME | 1.7 (0.79)
  12,13-EpOME | 0.96 (0.29)
  9,10-EpODE | 0.55 (0.54)
  12,13-EpODE | 0.12 (0.066)
  15,16-EpODE | 3.5 (3.4)
  9-KODE | 14 (6.3)
  13-KODE | 7.2 (3.8)
  12,13-Ep-9-KODE | 3.7 (2.8)
  5-KETE | 0.025 (0.019)
  LTB5 | 0.1 (0.094)
  10-Nitrooleate | 0.096 (0.054)
  10-Nitrolinoleate | 0.11 (0.069)
  PGE1 | 0.24 (0.15)
  PGE2 | 2.1 (1.8)
  PGF2a | 0.14 (0.14)
  15-deoxy PGJ2 | 0.033 (0.012)
  PGE3 | 0.13 (0.17)
  Sum TriHOMEs | 57 (56)
  PEA | 7.9 (6.8)
  SEA | 7.9 (6.7)
  OEA | 0.32 (0.38)
  LEA | 0.043 (0.035)
  aLEA | 0.0047 (0.0036)
  Dihomo GLA EA | 0.0022 (0.003)
  AEA | 0.019 (0.011)
  DEA | 0.17 (0.24)
  1-OG | 870 (1300)
  2-OG | 190 (270)
  1-LG | 300 (540)
  2-LG | 2.3 (1.1)
  1-AG | 14 (12)
  2-AG | 15 (30)
  NO-Gly | 0.48 (0.22)
  NA-Gly | 0.017 (0.02)
  C14 Ceramide | 1.4 (1.1)
  C16 Ceramide | 6.6 (4.7)
  C18 Ceramide | 1.2 (0.66)
  C20 Ceramide | 2 (1.4)
  C24 Ceramide | 5.7 (4.9)
  18:1 Sphingosine | 15 (8.9)

2. Primary Outcome: Volar Forearm Sweat Lipid Mediator Concentrations Following Exercise
Description: as for outcome 1
Time Frame: measured at study visit 1, detected lipid mediator concentrations reported
Population: Of the 14 subjects recruited for this study, only 7 provided usable data for this primary outcome.
Measure: Mean (Standard Deviation); unit: picomoles per milliliter
Arm/Group | Single Group
Number analyzed (Participants) | 7
picomoles per milliliter
  9-HODE | 2.4 (1.9)
  13-HODE | 5.2 (3.9)
  9-HOTrE | 0.6 (0.5)
  13-HOTrE | 1.5 (1.4)
  5-HETE | 0.023 (0.018)
  8-HETE | 0.14 (0.061)
  9-HETE | 0.029 (0.018)
  11-HETE | 0.012 (0.0061)
  12-HETE | 0.04 (0.031)
  15-HETE | 0.074 (0.054)
  12-HEPE | 0.029 (0.015)
  9,10-e-DiHO | 21 (12)
  9,10-DiHOME | 3.1 (1.8)
  12,13-DiHOME | 2.8 (1.6)
  9,10-DiHODE | 0.56 (0.68)
  12,13-DiHODE | 0.3 (0.12)
  15,16-DiHODE | 1.9 (2.3)
  5,6-DiHETrE | 0.026 (0.037)
  8,9-DiHETrE | 0.24 (0.25)
  11,12-DiHETrE | 0.022 (0.026)
  14,15-DiHETrE | 0.041 (0.018)
  9,10-EpOME | 0.46 (0.31)
  12,13-EpOME | 0.36 (0.22)
  9,10-EpODE | 0.19 (0.18)
  12,13-EpODE | 0.019 (0.014)
  15,16-EpODE | 0.82 (0.86)
  9-KODE | 1.5 (1.4)
  13-KODE | 0.89 (0.6)
  12,13-Ep-9-KODE | 3.4 (1.8)
  5-KETE | 0.02 (0.017)
  LTB5 | 0.099 (0.082)
  10-Nitrooleate | 0.074 (0.043)
  10-Nitrolinoleate | 0.087 (0.078)
  PGE1 | 0.85 (1)
  PGE2 | 1.1 (1.3)
  PGF2a | 0.44 (0.74)
  15-deoxy PGJ2 | 0.046 (0.036)
  PGE3 | 0.18 (0.21)
  Sum TriHOMEs | 130 (130)
  PEA | 14 (25)
  SEA | 15 (25)
  OEA | 0.11 (0.093)
  LEA | 0.019 (0.01)
  aLEA | 0.0033 (0.0024)
  Dihomo GLA EA | 0.0023 (0.0036)
  AEA | 0.017 (0.025)
  DEA | 0.015 (0.013)
  1-OG | 11 (14)
  2-OG | 7 (7.3)
  1-LG | 2.1 (1.8)
  2-LG | 0.34 (0.36)
  1-AG | 1.8 (3.1)
  2-AG | 0.79 (1)
  NO-Gly | 0.15 (0.13)
  NA-Gly | 0.01 (0.012)
  C14 Ceramide | 0.23 (0.18)
  C16 Ceramide | 1 (1)
  C18 Ceramide | 0.29 (0.34)
  C20 Ceramide | 0.36 (0.34)
  C24 Ceramide | 0.88 (0.8)
  18:1 Sphingosine | 4.9 (4.6)

3. Primary Outcome: Lower Back Sweat Lipid Mediator Concentrations Following Pilocarpine Stimulation
Description: as for outcome 1
Time Frame: measured at study visit 1, detected lipid mediator concentrations reported
Population: Of the 14 subjects recruited for this study, only 4 provided usable data for this primary outcome.
Measure: Mean (Standard Deviation); unit: picomoles per milliliter
Arm/Group | Single Group
Number analyzed (Participants) | 4
picomoles per milliliter
  9-HODE | 17 (11)
  13-HODE | 81 (42)
  9-HOTrE | 1.8 (0.65)
  13-HOTrE | 2.6 (1.1)
  5-HETE | 0.15 (0.1)
  8-HETE | 0.23 (0.21)
  9-HETE | 0.12 (0.083)
  11-HETE | 0.2 (0.27)
  12-HETE | 0.3 (0.22)
  15-HETE | 0.32 (0.2)
  12-HEPE | 0.15 (0.11)
  9,10-e-DiHO | 36 (13)
  9,10-DiHOME | 2.6 (0.73)
  12,13-DiHOME | 2.2 (0.52)
  9,10-DiHODE | 0.38 (0.16)
  12,13-DiHODE | 0.34 (0.14)
  15,16-DiHODE | 0.55 (0.16)
  5,6-DiHETrE | 2.8 (1.8)
  8,9-DiHETrE | 0.1 (0.22)
  11,12-DiHETrE | 0.28 (0.039)
  14,15-DiHETrE | 0.34 (0.067)
  9,10-EpOME | 1.6 (1.1)
  12,13-EpOME | 1.6 (1.3)
  9,10-EpODE | 0.28 (0.15)
  12,13-EpODE | 0.2 (0.1)
  15,16-EpODE | 0.49 (0.34)
  9-KODE | 11 (9.2)
  13-KODE | 6 (2.9)
  12,13-Ep-9-KODE | 2.6 (0.94)
  5-KETE | 0.1 (0.12)
  LTB5 | 0.13 (0.093)
  10-Nitrooleate | 0.75 (1.2)
  10-Nitrolinoleate | 0.26 (0.31)
  PGE1 | 0.11 (0.046)
  PGE2 | 0.62 (0.28)
  PGF2a | 0.27 (0.15)
  PGE3 | 0.17 (0.13)
  Sum TriHOMEs | 12 (11)
  PEA | 47 (65)
  SEA | 53 (73)
  OEA | 0.55 (0.46)
  LEA | 0.14 (0.14)
  aLEA | 0.11 (0.14)
  Dihomo GLA EA | 0.05 (0.083)
  AEA | 0.14 (0.19)
  DEA | 0.028 (0.069)
  1-OG | 300 (210)
  2-OG | 46 (47)
  1-LG | 110 (82)
  2-LG | 2.6 (1.3)
  1-AG | 10 (12)
  2-AG | 2.6 (1.3)
  NO-Gly | 0.25 (0.26)
  NA-Gly | 0.027 (0.057)
  C14 Ceramide | 0.49 (0.28)
  C16 Ceramide | 1.7 (1.6)
  C18 Ceramide | 0.34 (0.32)
  C20 Ceramide | 0.33 (0.26)
  C24 Ceramide | 0.41 (0.28)
  18:1 Sphingosine | 8.1 (12)

4. Primary Outcome: Anterior Distal Thigh Sweat Lipid Mediator Concentrations Following Pilocarpine Stimulation
Description: as for outcome 1
Time Frame: measured at study visit 2, detected lipid mediator concentrations reported
Population: Of the 14 subjects recruited for this study, only 4 provided usable data for this primary outcome.
Measure: Mean (Standard Deviation); unit: picomoles per milliliter
Arm/Group | Single Group
Number analyzed (Participants) | 4
picomoles per milliliter
  9-HODE | 19 (9.9)
  13-HODE | 48 (24)
  9-HOTrE | 1.8 (0.54)
  13-HOTrE | 5.2 (1)
  5-HETE | 0.067 (0.059)
  8-HETE | 0.17 (0.066)
  9-HETE | 0.12 (0.043)
  11-HETE | 0.12 (0.075)
  12-HETE | 0.31 (0.14)
  15-HETE | 0.26 (0.28)
  12-HEPE | 0.13 (0.057)
  9,10-e-DiHO | 35 (5.5)
  9,10-DiHOME | 2.9 (0.89)
  12,13-DiHOME | 2.4 (0.69)
  9,10-DiHODE | 0.46 (0.095)
  12,13-DiHODE | 0.7 (0.13)
  15,16-DiHODE | 0.99 (0.31)
  5,6-DiHETrE | 2.7 (1.2)
  8,9-DiHETrE | 0.62 (0.45)
  11,12-DiHETrE | 0.19 (0.072)
  14,15-DiHETrE | 0.19 (0.087)
  9,10-EpOME | 1.7 (0.54)
  12,13-EpOME | 1.6 (0.47)
  9,10-EpODE | 0.8 (0.66)
  12,13-EpODE | 0.25 (0.14)
  15,16-EpODE | 0.95 (0.45)
  9-KODE | 21 (17)
  13-KODE | 9.3 (7.3)
  12,13-Ep-9-KODE | 3.3 (1.4)
  5-KETE | 0.04 (0.018)
  LTB5 | 0.088 (0.068)
  10-Nitrooleate | 0.12 (0.14)
  10-Nitrolinoleate | 0.16 (0.019)
  PGE1 | 0.18 (0.15)
  PGE2 | 0.36 (0.38)
  PGF2a | 0.44 (0.45)
  PGE3 | 0.15 (0.14)
  Sum TriHOMEs | 36 (14)
  PEA | 18 (6.4)
  SEA | 18 (5.8)
  OEA | 0.31 (0.24)
  LEA | 0.078 (0.039)
  aLEA | 0.022 (0.005)
  Dihomo GLA EA | 0.00037 (0.0058)
  AEA | 0.013 (0.005)
  DEA | 0.053 (0.061)
  1-OG | 200 (88)
  2-OG | 37 (16)
  1-LG | 81 (41)
  2-LG | 2.1 (0.6)
  1-AG | 13 (5.4)
  2-AG | 4.2 (0.72)
  NO-Gly | 0.23 (0.14)
  NA-Gly | 0.02 (0.013)
  C14 Ceramide | 0.24 (0.15)
  C16 Ceramide | 1.5 (1.2)
  C18 Ceramide | 0.31 (0.25)
  C20 Ceramide | 0.36 (0.32)
  C24 Ceramide | 1 (0.99)
  18:1 Sphingosine | 2.2 (4.5)

5. Primary Outcome: Change in Plasma Lipid Mediator Concentrations Before and After Oral Ibuprofen Administration
Description: Approximately 100 lipid mediators will be measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Assayed lipid mediators include oxygenated lipids, endocannabinoids, and endocannabinoid-like molecules.
Time Frame: measured at four timepoints at study visit 4, detected lipid mediator concentrations for first timepoint reported
Population: Of the 14 subjects recruited for this study, only 9 provided usable data for this primary outcome.
Measure: Geometric Mean (Full Range); unit: picomoles per milliliter
Arm/Group | Single Group
Number analyzed (Participants) | 9
picomoles per milliliter
  PGE1 | 0.126 [0.04 to 0.421]
  PGE2 | 0.159 [0.06 to 0.6]
  PGF2a | 5.47 [1.43 to 23.7]
  13-HODE | 23 [11.7 to 40.7]
  9-HODE | 8.77 [5.38 to 16]
  13-HOTE | 1.56 [0.92 to 4.65]
  9-HOTE | 1.19 [0.71 to 2.43]
  15-HETE | 0.861 [0.14 to 3.56]
  12-HETE | 1.31 [0.66 to 6.38]
  11-HETE | 0.408 [0.2 to 0.88]
  5-HETE | 0.425 [0.02 to 1.86]
  17-HDoHE | 2.55 [0.1 to 34.7]
  9,10-e-DiHO | 10.4 [5.76 to 34.1]
  12,13-DiHOME | 4.13 [2.24 to 10.4]
  9,10-DiHOME | 4.44 [1.44 to 12]
  15,16-DiHODE | 15 [6.96 to 37.5]
  12,13-DiHODE | 1.77 [0.3 to 7.52]
  9,10-DiHODE | 0.458 [0.2 to 1.04]
  14,15-DiHETrE | 1.17 [0.7 to 2.77]
  11,12-DiHETrE | 1.11 [0.56 to 3.09]
  5,6-DiHETrE | 0.406 [0.06 to 1.04]
  17,18-DiHETE | 20.2 [7.4 to 33.2]
  19,20-DiHDoPA | 1.91 [0.76 to 4.13]
  Sum TriHOMEs | 7.88 [4.64 to 12.2]
  9(10)-EpO | 9.96 [2.37 to 45.8]
  12(13)-EpOME | 4.1 [1.14 to 11.8]
  9(10)-EpOME | 1.12 [0.26 to 4.7]
  15(16)-EpODE | 3.95 [0.95 to 11.3]
  9(10)-EpODE | 1.02 [0.35 to 10.2]
  13-KODE | 1.89 [0.13 to 19.3]
  9-KODE | 3.09 [0.67 to 15.7]
  OEA | 4.14 [2.83 to 8.65]
  LEA | 1.19 [0.67 to 1.95]
  aLEA | 0.0968 [0.04 to 0.29]
  Dihomo GLA EA | 0.168 [0.05 to 0.39]
  AEA | 0.627 [0.29 to 0.92]
  DEA | 0.298 [0.21 to 0.48]
  DHEA | 0.76 [0.28 to 1.46]
  NO-Gly | 3.5 [1.62 to 9.44]
  NA-Gly | 0.833 [0.34 to 1.63]
  OG | 393 [212 to 702]
  LG | 238 [67.6 to 820]
  AG | 20.7 [10 to 51.2]

6. Secondary Outcome: Change in Pilocarpine-stimulated Sweat Lipid Mediator Concentrations Before and After Oral Ibuprofen Administration
Description: as for outcome 5
Time Frame: measured at four timepoints at study visit 4, detected lipid mediator concentrations for first timepoint reported
Population: Of the 14 subjects recruited for this study, only 9 provided usable data for this primary outcome.
Measure: Geometric Mean (Full Range); unit: picomoles per milliliter
Arm/Group | Single Group
Number analyzed (Participants) | 9
picomoles per milliliter
  PGE1 | 0.453 [0.12 to 4.91]
  PGE2 | 2.71 [0.34 to 51.6]
  13-HODE | 21.9 [3.72 to 69.6]
  9-HODE | 7.72 [1.69 to 23.4]
  13-HOTE | 1.08 [0.29 to 3.23]
  9-HOTE | 1.08 [0.53 to 3.25]
  20-HETE | 0.742 [0.25 to 1.74]
  15-HETE | 0.311 [0.06 to 4.05]
  12-HETE | 0.965 [0.52 to 1.7]
  11-HETE | 0.0882 [0.01 to 0.39]
  8-HETE | 0.0618 [0.01 to 0.18]
  5-HETE | 0.138 [0.04 to 0.36]
  15-HEPE | 0.0576 [0.00136 to 0.3]
  12-HEPE | 0.0781 [0.01 to 0.23]
  17-HDoHE | 0.46 [0.09 to 7.41]
  9,10-e-DiHO | 58.4 [39 to 135]
  12,13-DiHOME | 1.89 [0.9 to 3.6]
  9,10-DiHOME | 3.61 [1.85 to 7.66]
  15,16-DiHODE | 1.49 [0.43 to 5.65]
  12,13-DiHODE | 0.332 [0.12 to 1.34]
  9,10-DiHODE | 0.35 [0.1 to 0.87]
  14,15-DiHETrE | 0.341 [0.09 to 1.09]
  11,12-DiHETrE | 0.231 [0.07 to 1.02]
  5,6-DiHETrE | 3.29 [1.28 to 10.7]
  17,18-DiHETE | 1.76 [0.31 to 6.72]
  Sum TriHOMEs | 31.7 [11.4 to 93.5]
  9(10)-EpO | 2.81 [0.89 to 6.54]
  12(13)-EpOME | 0.485 [0.08 to 1.31]
  9(10)-EpOME | 0.657 [0.16 to 1.93]
  15(16)-EpODE | 0.491 [0.04 to 4.5]
  12(13)-EpODE | 0.0703 [0.02 to 0.14]
  9(10)-EpODE | 0.194 [0.04 to 0.51]
  13-KODE | 2.17 [0.3 to 13.2]
  9-KODE | 5.35 [0.64 to 38.5]
  12(13)-Ep-9-KODE | 1.82 [0.72 to 3.64]
  10-Nitrooleate | 1.78 [0.36 to 6.24]
  9-Nitrooleate | 0.729 [0.09 to 3.76]
  10-Nitrolinoleate | 0.297 [0.16 to 0.6]
  OEA | 0.586 [0.09 to 2.7]
  LEA | 0.0447 [0.01 to 0.22]
  NO-Gly | 0.156 [0.01 to 0.55]
  NA-Gly | 0.0627 [0.01 to 0.23]
  OG | 61.5 [2.67 to 5620]
  LG | 4.11 [0.46 to 21.2]
  AG | 4.2 [0.15 to 836]

7. Secondary Outcome: Change in Plasma Ibuprofen Concentrations
Description: Plasma concentration of ibuprofen prior to and 30 min, 2 hr and 4 hr after oral administration
Time Frame: measured at four timepoints at study visit 4
Population: Of the 14 subjects recruited for this study, only 9 provided usable data for this primary outcome.
Measure: Geometric Mean (Full Range); unit: micrograms per milliliter
Arm/Group | Single Group
Number analyzed (Participants) | 9
micrograms per milliliter
  Prior to administration | 0 [0 to 0]
  30 min after administration | 18.8 [3.4 to 65.3]
  2 hr after administration | 48.3 [39.1 to 75.9]
  4 hr after administration | 33.8 [14.9 to 90.1]

8. Secondary Outcome: Change in Sweat Ibuprofen Concentrations
Description: Sweat concentration of ibuprofen prior to and 30 min, 2 hr and 4 hr after oral administration
Time Frame: measured at four timepoints at study visit 4
Population: Of the 14 subjects recruited for this study, only 9 provided usable data for this primary outcome.
Measure: Geometric Mean (Full Range); unit: micrograms per milliliter
Arm/Group | Single Group
Number analyzed (Participants) | 9
micrograms per milliliter
  Prior to administration | 0 [0 to 0]
  30 min after administration | 0 [0 to 0]
  2 hr after administration | 0 [0 to 0]
  4 hr after administration | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events collected from November 2016 to June 2017 (6 months)
Arm/Group | Single Group
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT02935894/Prot_000.pdf
  • Informed Consent Form (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02935894/ICF_001.pdf
  • Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT02935894/SAP_002.pdf